CLINICAL TRIAL: NCT03402373
Title: A 16-Week Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Nutritional Supplement Lycoderm on Its Impact on Skin Parameters in Healthy Female Subjects
Brief Title: Evaluation of the Nutritional Supplement Lycoderm on Its Impact on Skin Parameters
Acronym: Lycoderm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 4158LY0817
Record Dates: First submitted 2017-12-21; First posted 2018-01-18 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Skin Care

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind, Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycoderm (Experimental): soft gel contains nutritional supplement
  Interventions: Dietary Supplement: Lycoderm
- Placebo (Placebo Comparator): Soft gel without active ingredients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lycoderm — soft gel contains nutritional supplement
  Arms: Lycoderm
Dietary Supplement: Placebo — soft gel without active ingredients
  Arms: Placebo

SUMMARY:
Carotenoids and polyphenols are assumed to have an active role in skin health. Sources for these phytonutrient are fruits and vegetables. They are widely applied as skin protectants, and supplementation with carotenoids have shown to protect against erythema caused by UV-radiation. UV radiation generates reactive oxygen species in the skin, which induces cellular signaling that may impair cell cycle, cell growth, and regeneration or repair processes.

DETAILED DESCRIPTION:
The face holds an integral role in human social communication and how humans are perceived as attractive. In addition to structural facial features, studies have shown that skin appearance is highly weighed in the perception of beauty and is determined primarily by its coloration and surface topography. Aging is caused by two processes, intrinsic and extrinsic. The sun is the primary cause of extrinsic aging and has also been shown to alter the normal course of intrinsic or natural aging. On the molecular level, various hypotheses have been proposed to explain aging, with free radical theory being prominent. The free radical theory addresses the concept of intrinsic biological instability of living systems, in which free radicals and other reactive oxygen species (ROS) damage biomolecules, and this damage results in aging of the skin (as well as other systems).

The aim of this study is to examine the effects of an oral antioxidant supplement on skin aging and skin condition.

ELIGIBILITY:
Inclusion Criteria:

1. Females between ages of 35 and 55 years old, inclusive at enrollment
2. Subjects in good general health with no serious illnesses which might interfere with study participation per assessment of investigator.
3. Subjects with BMI <30 kg/m2
4. Nonsmokers (self-reported)
5. Agree to maintain current dietary regimen
6. Agree to maintain current cosmetic regimen
7. Skin Type II/ III.
8. Subjects with dull skin, lack of radiance, uneven skin tone, lines and wrinkles as determined by an expert grader at Baseline.

Exclusion Criteria:

1. Subjects with known allergies to soybeans, coconut, tomatoes, or rosemary.
2. Subjects that are not willing to to maintain current dietary regimen
3. Subjects that underwent extensive sunbathing in the month before study initiation or who plan to have excessive sun exposure or use a tanning bed/booth during the study.
4. Subjects that underwent procedures using injectables such as Botox or other fillers in 2 months before screening or who plan to undergo such procedures during the study.
5. Subjects with drastic change in body weight (greater than 10% 1 month prior to screening or during the study
6. Intake of vitamin or dietary supplements (especially Vitamin D3, carotenoids) during the month prior to screening
7. History of malabsorption diseases, liver diseases, or diseases of lipid metabolism.
8. History of photosensitizing disorders.
9. Use of medications which interact with the study procedures according to the principal investigator (during or prior to the study).
10. Subjects currently participating in a study or who have participated in any other clinical studies during the last 3 months prior to the study
11. Subjects having an acute or chronic disease or medical condition, including dermatological problems, which could put her at risk in the opinion of the Principal Investigator or compromise study outcomes.
12. History of allergic reactions, skin sensitization and/or known allergies to cosmetic ingredients, toiletries, sunscreens, etc.
13. Immunocompromised subjects .
14. Woman who started Hormone Replacement Therapy within the last three months preceding the screening visit.
15. Woman using oral contraception for less than three months before the screening visit or who has changed her contraceptive method within the three months before the Baseline visit or planning to modify her contraception treatment within the duration of the study.

17. Woman known to be pregnant, lactating or planning to become pregnant within six months. Subjects who become pregnant during the study must inform the Principal Investigator immediately and will be excluded from the study.

-

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Improves skin hydration | 16 weeks
  instrumental evaluation (Corneometer)
Improves skin smoothness and texture | 16 weeks
  image analysis (Antera)
Improves lines and wrinkles | 16 weeks
  image analysis (Clarity)
Improves skin barrier function | 16 weeks
  instrumental evaluation (VapoMeter)
Improves skin thickness and density | 16 weeks
  instrumental evaluation (DermaScan Ultrasound)
Increases dermal hemoglobin | 16 weeks
  instrumental evaluation (SIAScope).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frumento, Phd, Study Director — IRSI
Locations (1):
- International Research Services, Inc., Port Chester, New York, United States

IPD SHARING:
Plan to Share IPD: No